CLINICAL TRIAL: NCT01319708
Title: Mild Versus Conventional Ovarian Stimulation for Poor Responders Undergoing In Vitro Fertilisation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Siristatidis Charalampos, MD, PhD, Assistant Professor, Director of the ARU, National and Kapodistrian University of Athens
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1234561
Record Dates: First submitted 2011-03-08; First posted 2011-03-22 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-11

CONDITIONS: Infertility
Keywords: ovarian stimulation; climiphene citrate; Gonadotropin-Releasing Hormone agonists/antagonists; Follicle Stimulating Hormone
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- mild ovarian stimulation (Experimental): 100 mg CC by day 2 till 6, plus antagonist plus gonadotrophin 150-200IO until HCG triggering
  Interventions: Procedure: mild ovarian stimulation
- conventional ovarian stimulation (Active Comparator): 300-450 IU of FSH starting by day 2 of menstrual cycle together with a fixed dose of GnRH antagonist starting by day 6 till egg recovery, or same doses using a GnRH agonist long protocol
  Interventions: Procedure: conventional ovarian stimulation

INTERVENTIONS:
Procedure: mild ovarian stimulation — 100-150 mg of clomiphene citrate from day 2 till day 6 of the cycle and 150 mg of gonadotrophins as soon as 1 follicle is more than 14mm together with 1 fixed dose of GnRH antagonist until egg recovery
  Arms: mild ovarian stimulation
Procedure: conventional ovarian stimulation — 300-450 IU of FSH starting by day 2 of menstrual cycle together with a fixed dose of GnRH antagonist starting by day 6 till egg recovery, or same doses with GnRH agonist long protocol
  Arms: conventional ovarian stimulation

SUMMARY:
The investigators will examine the balance between IVF success in terms of outcome parameters, using a mild ovarian stimulation protocol, opposing it to the conventional stimulation regimens in poor responders undergoing IVF.

ELIGIBILITY:
Inclusion Criteria:

* poor responders (age>40, previous POR, abnormal OR test)
* indication for IVF
* regular cycling patients
* BMI 19-35

Exclusion Criteria:

* contraindication for clomiphene citrate use or to GnRH agonists antagonists
* BMI > 35

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2011-03; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
number of oocytes (COCs) | at oocyte recovery

SECONDARY OUTCOMES:
Number/rate of participants whom the IVF cycle was cancelled | After the 1st week of ovarian stimulation, no oocytes at OR
clinical pregnancy rate | 6 weeks
  Presence of fetal heart at transvaginal ultrasound at 6 weeks of gestation or 6 weeks after starting the intervention
live birth | more than 20 weeks
miscarriage | pregnancy loss before 20 weeks of gestation, after a positive pregnancy test
stimulation characteristics | from start of stimulation until embryo transfer
  total dose of gonadotropins administered,
cancellation rate | from start of stimulation until ET
  when premature ovulation was evident by the loss of follicle(s) prior to oocyte recovery, and in cases where there were no oocytes retrieved or no embryos produced for transfer and in failed fertilization

CONTACTS AND LOCATIONS:
Locations (1):
- 3rd Department of Obstetrics & Gynecology, Assisted Reproduction Unit, Athens, Chaidari, Greece